CLINICAL TRIAL: NCT03152292
Title: Management of Parkinson's Disease Psychosis in Actual Practice (The INSYTE Study)
Brief Title: The INSYTE (Management of Parkinson's Disease Psychosis in Actual Practice) Study
Status: Terminated | Type: Observational
Why Stopped: Study follow-up duration impacted by COVID-19pandemic and Sponsor terminated for business reasons
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ACP-NIS-001
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease Psychosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Parkinson Disease Psychosis (PDP) patients: PDP patients not treated with an antipsychotic at the time of enrollment
  Interventions: Other: Real-world, non-interventional
- Group 2: Parkinson Disease Psychosis (PDP) patients: PDP patients treated with an antipsychotic (other than NUPLAZID®) at the time of enrollment
  Interventions: Other: Real-world, non-interventional
- Group 3: Parkinson Disease Psychosis (PDP) patients: PDP patients treated with NUPLAZID® at the time of enrollment
  Interventions: Other: Real-world, non-interventional

INTERVENTIONS:
Other: Real-world, non-interventional — N/A - non-interventional

SUMMARY:
To examine the current disease progression of PDP, the clinical, economic, and humanistic impact of anti-psychotic therapy in the management of the condition in real-world settings, and the burden of the condition on patients and their caregivers

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females ≥ 18 with PDP
2. Ability to understand and read English
3. Patient is willing and able to sign an Informed Consent Form (ICF), or have a Legally Authorized Representative willing and able to consent on the patient's behalf
4. Possess the symptoms commonly associated with PDP, e.g., hallucinations and delusions that cannot be reasonably attributed to other causes

Exclusion Criteria:

1. Patient is unwilling to participate in the non-interventional study
2. Patient is currently participating in or is planning to participate in an investigational clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing hallucinations and delusions as a complication of Parkinson's Disease.
Sampling Method: Non-Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
The INSYTE (Management of Parkinson's Disease Psychosis in Actual Practice) | Approximately 36 months
  Describe the safety and effectiveness of antipsychotic therapies and other treatment approaches in the management of PDP. Describe comparative clinical, economic, and humanistic outcomes of treatment approaches for both patients and caregivers, in the context of real-world medical practice settings.

CONTACTS AND LOCATIONS:
Locations (69):
- United States (69):
  - North Central Neurology Associates, P.C., Cullman, Alabama
  - Peak Neurology and Sleep Medicine, LLC, Anchorage, Alaska
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Brain and Elective Spine Treatment Center, Laguna Hills, California
  - Silicon Valley Parkinson Center Inc., Los Gatos, California
  - Parkinson's Disease and Movement Disorder of Silicon Valley, Menlo Park, California
  - Jeri Yvonne Movement Disorders Neurology, Inc., Northridge, California
  - Pacific Movement Disorders Center, Santa Monica, California
  - Colorado Neurological Institute, Greenwood Village, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Neurology Offices of S. Florina, Boca Raton, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Inc., Boca Raton, Florida
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Intermed Medical Research Center, Miami, Florida
  - Ramon A. Gil, MD, PA, DBA Parkinson's Disease Treatment Center of SW Florida, Port Charlotte, Florida
  - NOVA Clinical Research, LLC, St. Petersburg, Florida
  - MS Center of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Southern Illinois Associates, LLC, Glen Carbon, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - American Health Network of Indiana, Avon, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Psychiatry Associates of Kansas City, Leawood, Kansas
  - Overland Park Surgical Specialties, LLC, Overland Park, Kansas
  - Southeast Neuroscience Center, Gray, Louisiana
  - LSU Health Sciences Center - New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - Parkinsons & Movement Disorders Center of Maryland, Elkridge, Maryland
  - Tufts Medical Center, Inc., Boston, Massachusetts
  - Neurology Center of New England, Foxborough, Massachusetts
  - University of Massachusetts, Worcester, Worcester, Massachusetts
  - Michigan State Neurology, East Lansing, Michigan
  - The Parkinson's and Movement Disorder Center, Farmington Hills, Michigan
  - Cornelius Robens, MD, PLLC, Traverse City, Michigan
  - Henry Ford Health System, West Bloomfield, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Neurology Consultants of Nebraska, Omaha, Nebraska
  - Las Vegas Neurology Center, Las Vegas, Nevada
  - Neurology Center of Las Vegas, Las Vegas, Nevada
  - The Cooper Health System, Camden, New Jersey
  - JFK Neuroscience Institute, Edison, New Jersey
  - Rutgers, Robert Wood Johnson, New Brunswick, New Jersey
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - University of Rochester Neurology, Rochester, New York
  - Alpha Neurology PC, Staten Island, New York
  - New York Medical College, Valhalla, New York
  - Excel Psychiatric Associates, Huntersville, North Carolina
  - Raleigh Neurology Associates, PA, Raleigh, North Carolina
  - Neurology and Neuroscience Associates, Inc., Akron, Ohio
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Renga A. Pakeeree, MD, Cuyahoga Falls, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Allegheny-Singer Research Institute, East Providence, Rhode Island
  - Jacinto Medical Group, Baytown, Texas
  - North Texas Movement Disorders Institute, Bedford, Texas
  - Texas Institute for Neurological Disorders (Texoma Neurology), Sherman, Texas
  - East Texas Medical Center Healthcare Associates, Tyler, Texas
  - CHRISTUS Trinity Frances Neuroscience Institute, Tyler, Texas
  - Medical Faculty Associates, Inc., Arlington, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Blacksburg Neurology, PC, Christiansburg, Virginia
  - Neurology Specialists, Norfolk, Virginia
  - Henrico Doctors' Neurology Associates LLC, Richmond, Virginia
  - Cascade Surgery Associates, PLLC DBA Northwest Neurology Electrodiagnostic Center, Auburn, Washington
  - Inland Northwest Research, LLC, Spokane, Washington
  - Vaught Neurological Services, PLLC, Beckley, West Virginia
  - Gundersen Lutheran Medical Center, Inc., La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No